Title:Study of the Effects Caloric Restriction and Exercise Training in Patients With Heart Failure and a Normal Ejection Fraction

NCT: NCT02636439 Date: 5/31/2019



Department of Internal Medicine/Section Cardiology

# SECRET-II, EFFECTS OF CALORIC RESTRICTION AND EXERCISE TRAINING IN PATIENTS WITH HEART FAILURE AND A NORMAL EJECTION FRACTION.

Informed Consent Form to Participate in Research Dalane Kitzman, MD, Principal Investigator

#### INTRODUCTION

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you have symptoms compatible with a disorder called heart failure with a normal ejection fraction. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to study the long-term effects of a weight loss and exercise program compared to a weight loss, exercise and strength training program on physical function, quality of life, and body composition.

HOW MANY PEOPLE WILL TAKE PART IN THE STUDY? Up to 90 people at this research site will take part in this study.

#### WHAT IS INVOLVED IN THE STUDY?

Screening Visit:

If you agree to take part in this study, you will come to the Clinical Research Unit (CRU) for an initial screening visit to have the following tests and procedures:

- Brief history and physical exam
- Echocardiogram and Doppler. This is a sound wave test (ultrasound) of your heart, arm, leg and/or neck performed while you are lying comfortably on a padded table. Harmless sound waves will be used to create images of your heart, neck, arm and/or leg. During the ultrasound test you will have a blood pressure cuff inflated around your arm and/or leg so we can check your blood pressure during the test. There are no known risks involved in the use of ultrasound. This test will take about 30 minutes.

 Adult Consent Form



- Measurements of your blood pressure, height and weight
- Meet with a registered dietician for nutritional assessment and review of diet history.
- A pulmonary function test (a harmless breathing test to check your lung function) may be performed.

This initial screening visit will take approximately 1 ½- 2 hours to complete.

#### Baseline Visits, BV1, BV2 and BV3:

If you are eligible and wish to continue, you will be asked to return to the Medical Center for the following testing and procedures. In order to participate in the study, you are not required to undergo all the tests and procedures, however, certain measures are required to assess eligibility. The CMP, comprehensive metabolic panel, is used as a broad screening tool to evaluate organ function and check for various medical conditions. CBC, complete blood count, is used to check for anemia. These blood tests must be obtained prior to study randomization. Your participation in the study will not be affected if you choose to not participate in one or more of the tests/procedures. Not all of these tests can be done in the same day. We will schedule a maximum of four baseline appointments at your convenience over a 3-4 week period.

- 1. Blood draw: About 93 cc (about six and a half tablespoons) of blood will be drawn from a vein in your arm. The total amount of blood withdrawn during the study will be approximately 186 cc. About 60 cc (about four tablespoons) will be used to measure your kidney hormone levels and other hormones that affect the heart.

  As part of this study, a blood sample will be obtained and DNA from your blood sample will be purified. DNA, or deoxyribonucleic acid, stores and transmits inherited traits, such as eye color or blood type. As part of this research project, your DNA will be studied in an effort to find out if there are genes that contribute to medical conditions
  - traits, such as eye color or blood type. As part of this research project, your DNA will be studied in an effort to find out if there are genes that contribute to medical conditions that are part of this study. Because we do not know how the results of this DNA study relate to your individual health, the results of the research will not be given to you or your doctor without your permission. These results will also not be placed in your medical records.
- 2. 6 minute walk test: You will be asked to walk at a brisk walking pace for six minutes at the Wake Forest University Clinical Research Center. The distance you cover will be recorded. During the walking test, there is a chance you could lose your balance, trip, or fall. To minimize this risk, we will make sure you have a clear walking path and that trained staff is always nearby.
- 3. Exercise test: You will be asked to walk on a treadmill while breathing through a mouthpiece or face mask, to measure your breathing. Your heart rate, rhythm, and blood pressure will also be monitored. The speed and grade will gradually increase making it harder for you to walk. Continue walking until you are short of breath or very tired and unable to continue. There is a small chance that the exercise test could lead to symptoms of heart disease or to injury. However, this will be minimized by the history




and physical examination beforehand, and the continual safety monitoring during the exercise test. The exercise test will be supervised by medical personnel trained to deal with any complications. This test will take about 40 minutes.

- 4. 2-Magnetic Resonance Imaging (MRI) scans: The MRI uses a strong magnet instead of x-ray energy to take electronic pictures. During the scan, you will lie on your back on a bed that will slowly glide into the MRI machine. The scanner makes loud noises, but you will wear headphones with built-in ear plugs to protect your ears. The first scan will take pictures of your heart, abdomen and/or the arteries in your arm or leg. You may be asked to do light exercise right before or during your MRI scan. During the MRI scan you will have a blood pressure cuff inflated around your arm and/or leg so we can take your blood pressure. The purpose of the MRI scan is to assess body composition (how much fat, bone, and muscle you have) and cardiac function. The second MRI scan will be of your head and brain. For part of this scan, you may be asked to wear a mask that will be attached to a machine called a RespirAct. This device is designed to maintain your oxygen (O2) levels while increasing your carbon dioxide (CO2) level slightly. The result of the increased CO2 is that the blood vessels in your brain will dilate allowing us to better understand how blood flows through your brain. While you may feel short of breath, you will not be deprived of oxygen at any point during the test. MRI scanners have been in clinical use for about 20 years. The MRI scanner uses a magnetic field and radio waves, not x-rays or other forms of radiation. To the best of our knowledge, there is no risk to having an MRI scan. Because strong magnetic fields are used for scanning, patients with inserted devices or objects known to be sensitive to strong magnetic fields (i.e. metallic foreign bodies inside your head or in your eyes, incompatible medical implants, pacemakers, brain stimulators, blood vessel clips, etc.) will not be allowed to participate in the MRI scan. The inside of the scanner is small. Some people feel nervous or anxious in such tight spaces. You will be able to stop the scan if you have these feelings. Each test will take about one hour.
- 5. Muscle biopsy: The skin of one of your thighs will be thoroughly cleaned and a local anesthetic (numbing medicine similar to what a dentist uses) will be used to numb your skin first and then your thigh muscle. After the numbing medicine takes effect, a very small incision (1/4 inch long) will be made in the skin of your thigh. A needle will be inserted multiple times to remove a small piece of muscle (about the size of a small pea). After the needle is removed, the doctor will apply pressure to your leg to prevent bleeding into the tissue and will close the incision with small pieces of sterile tape. This muscle sample will be studied to measure factors affecting muscle function, strength, endurance, and metabolism. This procedure takes about one hour to complete. To reduce the chance of bleeding, you cannot take aspirin, certain other pain relievers (like ibuprofen, Motrin<sup>TM</sup>, Advil<sup>TM</sup>, Aleve<sup>TM</sup>) or other medications that may affect bleeding, platelets, or bruising for 1 week before and for 3 days after the procedure. It is OK to use acetaminophen (Tylenol<sup>TM</sup> or Extra-strength Tylenol<sup>TM</sup>). You will also be asked to avoid strenuous physical activity for 36 hours before and after the procedure. You will be asked to fast (nothing to eat or drink except water for 12 hours before your visit). snack will be provided after the sampling. The numbing medicine injected into your




muscle will reduce the discomfort felt during removal of the small muscle sample. Temporary numbness of the skin near the sampling site can rarely occur, and very rarely, the numbness can persist. Bruising can occur. You may feel pain or soreness in the area of the sampling after the local anesthetic wears off. There is a slight risk of bleeding into the tissue and infection, however, pressure is applied to stop the bleeding and this procedure is done under sterile conditions to protect against infection. You will be given instructions on how to care for the incision and treat any pain or discomfort before you leave the clinic. A very small scar (1/4 inch) may develop. If you are allergic to the local anesthetic, you may experience dizziness, anxiousness, numbness of the lips and tightness of the throat. Medications to treat your reaction are kept close by if needed. If you are allergic or sensitive to adhesive tape, you may experience skin irritation or a rash where the tape was applied. These reactions go away within a short time. This test will take about one hour.

- 6. Dual X-ray Absorptiometry Scan: A DXA scan is a type of x-ray that measures your body composition (how much fat, bone and muscle you have) and your bone density. You will lie on a padded bed while the scanner moves over your body. This is a painless procedure that involves very low dose radiation. The purpose of the DXA scan is to assess the effects of the weight loss intervention. This may be seen in changes in bone density or body composition. The DXA scan involves exposure to radiation. The risk of this procedure is small and is similar to that received from clinical x-ray and nuclear medicine studies. The amount of radiation exposure that you will receive from this procedure is equivalent to a uniform whole body exposure of 4 millirem. This is equal to 0.01 times the amount of background radiation that the average person in the United States receives each year (annual background =300 millirem). This test will take about 30 minutes.
- 7. Muscle strength: Maximal isokinetic knee extensor strength will be measured via an isokinetic dynamometer (Biodex) at speeds of 60° and 180° per second with the participant sitting and the hips and knee flexed at 90°. All testing will be performed on both legs unless there is a reason not to test one of them, e.g., acute injury. To stabilize the hip joint and the trunk, subjects will be restrained with straps at the level of the chest, hip and thigh. Seat height and depth, as well as length of the lower leg, will be recorded to establish consistency between all tests. During testing, the lever arm will be 2 cm proximal to the anterior ankle crease. The knee joint center (lateral femoral condyle) will be aligned with the axis of rotation of the dynamometer. Start and stop angles will be set at 90° and 30°, respectively. Participants will be asked to extend and flex the knee and push as hard as possible against the resistance pad. Strength is assessed as peak torque and expressed in Newton-meters (Nm). The best performance of 2 trials will be selected for each side, and the averages of the left and right leg will be used in analyses. This test takes about 30 minutes.
- 8. Resting Metabolism Assessment: You will be asked to lie flat in a dimly lit room for up to 45 minutes while breathing into a special mask to measure your metabolism. Based on your breathing measures, the study staff will be able to calculate your resting

 Adult Consent Form



metabolism. This information will be used to establish a safe and effective diet plan. This is a non-invasive test; however, some participants do have the feeling of claustrophobia during the test. This test takes about one hour.

- 9. Health Related Quality of Life: You will be asked to complete a questionnaire of your physical symptoms, daily activities, mood, and support from friends and family.
- 10. Cognitive testing: You will be given tests of memory and thinking, and asked questions about daily functioning, mood, and other behaviors. Some of the tests will be completed with the use of a computer or tablet, while other tests will require the use of paper and pencil.
- 11. Physical Performance Battery: You will be asked to undergo physical function assessments including testing your hand grip strength. You will also be asked to do everyday tasks such as standing from a chair, balance while standing and a 4 meter walk test.
- 12. Physical Activity Monitoring: We will ask you to wear 2 small activity monitors for 1 week at the beginning and end of the study. One activity monitor will be worn on the wrist of your non-dominant hand, while the other will be worn on your right hip. You will wear the wrist activity monitor continuously, except when showering/bathing. The hip monitor will be removed for sleep, as well as showering and bathing. The monitor will collect data corresponding to the frequency, intensity, and duration of any physical activity you participate in. The wrist monitor will additionally track the quality and quantity of your sleep. The data will not be associated with your name or other personally identifying information; you will be assigned a study identification number.
- 13. Stool Sample: You will be asked to provide a stool sample for microbiome testing. Microbiome is the collection of microorganisms (such as bacteria, fungi, and viruses) that live in or on the human body. You will be provided instructions and a kit for collection.
- 14. COSMED K5: You may be asked to wear the COSMED K5 mask during 2 exercise intervention visits. One at the beginning of the 20 week sessions and one at the end.

All study outcome measures will be repeated at the end of the study, with the exception of the resting metabolic assessment.

After you have completed the entire study, you may be asked to return for a long-term follow-up visit. This will occur no earlier than 8 months post intervention and may be up to 4 years post intervention. The long-term follow-up visit will be conducted to assess changes in:

1-weight,

2-waist/hip ratio

3-exercise test,

4-SPPB, 5-grip strength and 6-minute walk for physical function,

 Adult Consent Form

| Version: | | | | |
|----------|---------|---------|-------|----|
| IRB Te | emplate | Version | 9.24. | 14 |



7-KCCQ (quality of life questionnaire)

8-DXA and MRI for body composition.

9-blood sample-inflammation markers, and gut hormones.

10-stool sample.

11-physical activity monitoring.

The "long-term visit" may be completed in 1 or 2 visits.

You may refuse to participate in one or more of these procedures and still participate in other study procedures without consequence.

We can send copies of your test results to your personal physician. Even if you do not wish to have any of your medical information sent to your physician, you can still participate in this research study.

Do you request that we send important medical findings from your study tests/exams to your personal physician?

| [ ] Yes | [ ] No | Initials |
|---------|--------|----------|

#### Randomization:

After completing these baseline tests, you will be randomized into one of the 2 study groups described below and then asked to repeat the same tests after 20 weeks. Randomization means that you are put into a group by chance. It is like flipping a coin. You will have an equal chance of being placed in either group.

#### Diet and Exercise Only Group:

This group will participate in a calorie restrictive diet with a goal of losing 1 pound per week throughout the study. Two meals and one snack will be provided for subjects participating in this part of the study. Options and suggestions will be given for breakfast since this meal will not be provided. The amount and type of food will be determined based on your age, gender, and measures of resting metabolism. Diets will be individually designed to promote weight loss by reducing calories by 300-400 calories per day. If assigned to this group you will be asked to pick up meals prepared especially for you from the CRU three days per week throughout the duration of the study.

The exercise program will consist of walking or cycling. Your exercise program will be designed specifically for you based on your heart rate. The exercise program will take place at Wake Forest University Clinical Research Center and will be supervised. If you are assigned to participate in this part of the study, you will be asked to exercise three days per week throughout the entire study.

#### Diet, Exercise and Strength Training:

This group will participate in the above mentioned diet and exercise with the addition of strength training added to the exercise portion. Strength training is a type of physical exercise specializing

 Adult Consent Form

| Version: | | | |
|----------|-----------------|------|----|
| IRB Te | emplate Version | 9 24 | 14 |



in the use of resistance to induce muscular contraction which builds the strength, anaerobic endurance, and size of skeletal muscles. If you are randomized to this group, you will have a short rest period before initiating the resistance training (RT) session.

## Storage of Biological Tissue

If you agree to participate in this study, we will draw 20 cc's (about two tablespoons) of blood to be used for future research. A sample of muscle tissue may also be saved for future research. These samples will be kept and may be used in future research to learn more about other diseases. Your samples will be obtained in the CRU at Wake Forest University Baptist Medical Center.

The samples will be stored in the CRU and will be given only to researchers approved by Dr. Dalane Kitzman. An Institutional Review Board (IRB) must also approve any future research study using your samples.

Your blood/tissue samples will be stored de-identified, which means that no identifying information will be stored with it. Researchers will not know the name, date of birth, medical record number, social security number, etc., of the person who donated the samples.

The research that may be performed with your blood/tissue samples is not designed to help you

The research that may be performed with your blood/tissue samples is not designed to help you specifically. There is no personal benefit to you from taking part in this aspect of the research study. It might help people who have diseases at some point in the future, but it is not known if this will happen. The results of the research performed with your blood/tissue will not be given to you or your doctor. The results will not be put in your medical record. The research using your blood/tissue samples will not affect your care.

Your blood/tissue samples will be used only for research and will not be sold. The findings from this research may result in the future development of products that are of commercial value. There are no plans to share any of the profits with you which may occur as a result of the research.

In the future, people who do research may need to know more about your health. While the study investigator may give reports about your health, he/she will NOT be given your name, address, phone number, or any other identifying information about who you are, unless you agree to be contacted in the future.

| YES you may contact for future research | ch studies |
|-----------------------------------------|-------------------------------|
| NO I do not want to be contacted regard | ding future research studies. |

#### HOW LONG WILL I BE IN THE STUDY?

You will be in the study for about 20 weeks plus the time required for baseline visits (3-4 weeks).

You can stop participating at any time. If you decide to stop participating in the study, we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences.


Adult Consent Form



Being in this study involves some risk to you. You should discuss the risk of being in this study with the study staff. Risks and side effects related to the procedures we are studying include:

Blood draw- You may experience discomfort, bruising and/or bleeding where the needle is inserted. Occasionally some people become dizzy lightheaded or feel faint. Infection may occur on rare occasions. Frequent donation of blood can result in low iron in your blood (iron deficient anemia).

Exercise and Resistance Training Program- Blood pressure and heart rate will be measured and recorded before each exercise session. The risks of the exercise and program are minimal but may include fainting, dizziness, irregular heartbeat, chest pain, heart attack, or extremely rarely, sudden death, and stresses and strains of muscles, twisted ankles, or falls. All exercise classes will be closely supervised by exercise technicians, who will instruct subjects in proper exercise techniques. If you are diabetic, you may be at an increased risk for hypoglycemia, a drop in your blood sugar. The symptoms of hypoglycemia may vary from person to person. Some of the most common are: confusion, dizziness, feeling shaky, hunger, headaches, pounding heart, racing pulse, weakness and trembling.

MRI Scan - The MRI scan is painless, and there are known no risks associated with the test. The MRI scans are being conducted only for the purpose of research. They are different than what is used in the clinical setting to detect or discover medical conditions. This is not a substitute for a clinical MRI scan. Research personnel will analyze the scans only for the specified research findings. If we should happen to see an abnormal finding that may be harmful to your health, we will notify you and your personal physician if you ask us to. Unexpected findings on the limited research scan will occasionally allow early discovery of a medical condition for which you may need treatment. They may also cause undue worry or result in additional testing, sometimes costly, which may or may not benefit your health.

RespirAct-(used during your brain MRI)- The RespirAct has been used in over 1000 studies and has been carefully evaluated for safety. Risks associated with the RespirAct procedure may include slight elevation in blood pressure (about 10mmHg), feeling short of breath or lightheaded, and headaches. We will monitor your heart rate and blood pressure during the test. You will be given an emergency signal for the duration of the MRI scan. You may use this signal to stop the RespirAct or the MRI scan at any time.

Dietary Intervention- There is no risk associated with measuring dietary intake or of eating a prepared diet to lose weight. Changes in usual bowel function (diarrhea and/or constipation) may occur when beginning dietary intervention due to differences between the SECRET-II diet and your usual diet. Under conditions of rapid weight loss (more than 5 pounds per week), there is a very small chance of developing gall bladder disease.

 Adult Consent Form



If you are a diabetic, you may be at an increased risk for hypoglycemia, a drop in your blood sugar. Please notify the study staff if you experience any hypoglycemic episodes.

There is also a risk of illness from improperly handled food. The CRU metabolic kitchen maintains strict policies and procedures to ensure food safety, but you will also need to handle food safely and as instructed to minimize risk.

In addition, there is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. There also may be other side effects that we cannot predict. You should tell the research staff about all the medications, vitamins and supplements you take and any medical conditions you have. This may help avoid side effects, interactions and other risks.

If you participate in this study, you will be exposed to amounts of radiation above what you would normally receive in daily life. To be sure that you do not receive an unhealthy amount of radiation from your participation in this study, you should let your study doctor know if you have had, or are going to have, any other scans or x-rays as part of your medical or dental care. It is very important that you let your study doctor know if you already are participating in, or plan to participate in, any other research study that involves radiation exposure.

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure

And allowing only authorized people to have access to research records, will be made to keep your information safe.

A Data Safety and Monitoring Committee, an independent group of experts, will be reviewing the data from this research throughout the study.

Pregnant women are excluded from participation in this study.

## ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct benefit to you. A possible benefit is that by losing weight and/or increasing your physical activity you may reduce your risk for diabetes and heart disease, and you may increase your fitness. The testing procedures may also detect other disorders previously unknown to you. If successful, the information learned from this study will benefit other people in the future.

#### WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have.

## What About My Health Information?

In this research study, any new information we collect from you about your health or behaviors is considered Protected Health Information. The information we will collect for this research

 Adult Consent Form

| Version: | | | | |
|----------|--------|---------|------|----|
| IRB Te | mplate | Version | 9 24 | 14 |



study includes: Information that identifies you, but is not limited to, such things as your name, address, telephone number, and date of birth. Your personal health information includes all information about you which is collected or created during the study for research purposes. It also includes your personal health information that is related to this study and that is maintained in your medical records at this institution and at other places such as other hospitals and clinics where you may have received medical care. Examples of your personal health information include your health history, your family health history, how you respond to study activities or procedures, laboratory and other test results, medical images, photographs/videotapes/audiotapes and information from study visits, phone calls, surveys, and physical examinations.

We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer. Only the following people or organizations will be granted access to your Protected Health Information:

- 1) The study investigator and his/her staff, or others at Wake Forest University Health Sciences who oversee research
- 2) Other people or laboratories providing services for this research project on behalf of Wake Forest University Health Sciences and Wake Forest University Baptist Medical Center.
- 3) Monitors, auditors, IRB or other regulatory agencies will be granted direct access to the participant's original medical record for verification of clinical trial procedures or data, without violating confidentiality of the participant and to the extent permitted by other applicable laws.
- 4) FDA and NIH/NIA

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study is maintained in the research records. Any research information entered into your medical record will be kept for as long as your medical record is kept by the Medical Center. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell Dr. Dalane W. Kitzman that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:

 Adult Consent Form



#### Dr. Dalane W. Kitzman

However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Laboratory test results and other medical reports created as a result of your participation in the research study may be entered into the computer systems of Wake Forest University Health Sciences and North Carolina Baptist Hospital. These will be kept secure, with access to this information limited to individuals with proper authority, but who may not be directly involved with this research study.

A North Carolina Baptist Hospital (NCBH) medical record will be created for all study participants. Information about your participation in the study will be placed in the NCBH medical record, along with any routine medical test results that were obtained at NCBH as part of this study.

If you withdraw your authorization you will not be able to be in this study. If you withdraw your authorization, no new health information that identifies you will be gathered after that date. Your health information that has already been gathered may still be used and disclosed to others. This would be done if it were necessary for the research to be reliable. You will not have access to your health information that is included in the research study records until the end of the study. This authorization is valid for six years or five years after the completion of the study, whichever is longer.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health

 Adult Consent Form



Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

#### WHAT ARE THE COSTS?

There are no costs to you for taking part in this study. All the study costs, including the testing procedures, the exercise sessions, and the meals will be paid for by the study. Costs for your regular medical care, which are not related to this study, will be your own responsibility

#### WILL YOU BE PAID FOR PARTICIPATING?

You will be paid \$350 if you complete all the scheduled study visits. If you withdraw for any reason from the study before completion you will be paid \$50 for each completed study visit. If you participate in the long-term follow up visit, you may receive up to \$100 for completion of all testing.

To receive payment, you must provide your social security number, name and address so that we can comply with IRS (Internal Revenue Service) reporting requirements. When payments are reported to the IRS, we do not let them know what the payment is for, only that you have been paid. If you do not wish to provide this information you can still take part in this study but you will not be paid.

## WHO IS SPONSORING THIS STUDY?

This study is being sponsored by the National Institutes of Health. The sponsor is providing money or other support to Wake Forest University Health Sciences to help conduct this study.

The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

## WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

Should you experience a physical injury or illness as a direct result of your participation in this study, Wake Forest University School of Medicine maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of such injuries or illnesses. To the extent research insurance coverage is available under this policy the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. Wake Forest University Baptist Medical Center holds the insurance policy for this coverage. It provides a maximum of \$25,000 coverage for each claim and is limited to a total of \$250,000 for all claims in any one year. The Wake Forest University School of Medicine, and the North Carolina Baptist Hospitals, Incorporated do not assume responsibility to pay for these medical services or to provide any other compensation for such injury or illness. Additional information may be obtained from the Medical Center's Director of Risk and Insurance Management, at

If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a

 Adult Consent Form

| Version: | |
|---------------------------|----|
| IRB Template Version 9 24 | 14 |



government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Dr. Kitzman at hours emergency, you may call the hospital operator at and ask to speak to the Cardiology Fellow on call.

#### WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest, your condition worsened, new information becomes available, you had an unexpected reaction, you failed to follow instructions, or because the entire study has been stopped.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Dalane W. Kitzman at operator at and ask to speak to the Cardiology Fellow on call.

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, you should contact the Chairman of the IRB at

You will be given a signed copy of this consent form.




## **SIGNATURES**

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Subject Name (Printed) | | | |
|---------------------------------|-------|----------|-------|
| Subject Signature | | Date/Tim | e |
| Person Obtaining Consent | | Date/Tim | e |
| Legal Representative Signature: | Date: | Time: | am pm |
